CLINICAL TRIAL: NCT00507260
Title: A Pilot Study to Evaluate a Nutritional Assessment Intervention to Improve Cancer-Related Fatigue Among Post-Allogeneic Blood and Marrow Transplantation Recipients
Brief Title: Nutritional Assessment Intervention to Improve Cancer-Related Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0515
Record Dates: First submitted 2007-07-24; First posted 2007-07-26 (Estimated); Last update posted 2014-12-24 (Estimated); Status verified 2014-12

CONDITIONS: Leukemia; Lymphoma; Fatigue
Keywords: Leukemia; Lymphoma; Post-Allogeneic Blood and Marrow Transplantation; Blood and Marrow Transplantation; BMT; Cancer-Related Fatigue; Fatigue; Nutritional Assessment; Nutritional Intervention; Malnutrition
MeSH Terms: conditions — Leukemia; Lymphoma; Fatigue; Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (Experimental): Control Group (Food Record)
  Interventions: Behavioral: Food Record
- Treatment Group (Experimental): Treatment Group (Food Record + Nutritional Consults)
  Interventions: Behavioral: Food Record; Other: Nutritional Consults

INTERVENTIONS:
Behavioral: Food Record — A record of the amount and kind of food and drink you intake will be completed.
Other: Nutritional Consults — Meeting with a dietician consultant regarding issues related to food intake. Participants will also receive the results from the food records.
  Arms: Treatment Group

SUMMARY:
Primary Objective:

1. To use the results from this pilot study to estimate the effect size of the nutritional intervention on fatigue and caloric intake.

Secondary Objectives:

1. To apply nutritional assessment tools for early detection of patients at risk for malnutrition.
2. To examine the feasibility of conducting this intervention study.
3. To describe cancer-related fatigue patterns among BMT patients at multiple time points during ambulatory visits.
4. To evaluate the effects of a nutritional intervention for post-allogeneic BMT recipients on adequacy of caloric intake in order to improve cancer-related fatigue scores.

DETAILED DESCRIPTION:
Recipients of an allogeneic BMT often experience fatigue as a side effect due to several factors, including high-dose chemotherapy and/or radiation therapy as well as stress from everyday activities that increase fatigue. In addition, after transplantation, the patient's ability to maintain regular nutritional needs (usually due to the unique diet that is required to help increase marrow function) is affected, which further increases fatigue levels. Researchers want to use information learned in this study to find out if nutritional intervention can help decrease fatigue levels and increase caloric intake.

Participating in this study involves routine visits to M. D. Anderson at the ambulatory treatment center. Before you can start on this study, you will be asked about any allergies you may have. You will also be asked some questions about your caregivers, such as how many caregivers you have, whether your caregiver will be able to attend the nutrition class with you, and whether the caregiver will record the food intake information. You will be asked these questions to help the study researcher decide if you are eligible to take part in this study. It should take about 30 minutes to collect this data. Your caregiver will be present while this data is being collected. You will be asked to fill out questionnaires about your medical history, personal demographics (such as your name, age, race, and gender), and fatigue levels. These questionnaires should take about less than 1 hour to complete. The study researcher will collect these questionnaires and put them in an envelope with a code ID number on the front cover, instead of your name or other personal information.

A dietitian will then set-up an appointment (within 3 days after your first visit to the ambulatory clinics) for a baseline test called indirect calorimetry. This test will be performed in your treatment room in the ambulatory treatment clinic to find out how many calories you need to have on a daily basis. For this test, you will be asked to sit quietly in your treatment room and breathe through a mouth piece with a nose clip on your nose for 10 minutes. This test will use a machine to collect the air that you breathe in (inhalation) and out (exhalation). The machine will use the information from your breathing to calculate how many calories you will need to intake each day. This entire process should take about 1 hour to complete. You will be given recommended levels of dietary caloric intake and your schedule for study activities within the first week of enrolling in this study. After this test, you will be randomized (as in the toss of a coin) to a group.

There will be 2 groups in this study. There will be about 6 participants in each group. If you are found to be eligible and you agree to take part in this study, you will be asked to draw a sealed envelope from a bag, which will show which study group you will be in. You will be allowed to draw only 1 envelope from the bag. You will have an equal chance of being assigned to either group.

Participants in 1 group will be given standard care (for the next 42 days) for allogeneic BMT at the ambulatory center. Participants in the other group will be given standard care (for the next 45 days) for allogeneic BMT at the ambulatory center as well as nutritional assessment and intervention. If your envelope has a label that says "standard," you will receive standard care only. If your envelope has a label that says "intervention," you will receive standard care as well as nutritional assessment and intervention.

During the first week on this study, you and your caregiver will receive training from the dietitian about putting information in a food record, which will include your name and the amount and kind of food and drink you intake from the time you get out of bed to the time you go to bed. On Days 7, 21, and 35 (Weeks 1, 3, and 5), the study researcher will remind you and your caregiver to start this food record and give you the recording sheets. You have to turn in 3 daily food records for the specified weeks. If you have some days off from the ambulatory center visits during that week, the study researcher would like you to complete a one-day food record on your day off as part of the 3 daily records.

If you have a different caregiver on any one of the weeks, the dietitian will train the new caregiver to record food and drinks on these days. The study researcher will collect the food records and give you a fatigue questionnaire on Days 14, 28, and 42. It should take about 30 minutes to complete. If you are not scheduled for a clinic visit on these specified days, the study researcher will meet with you on the first visit following these dates.

If you are in the standard care group, you will receive an indirect calorimetry test at the beginning of study, and you will submit 3-day food records every 2 weeks. You will not receive the results from these food records. Your health care provider may refer you to see a dietitian at any time during this study as part of your standard care. If at any time your caloric intake is considered to be 50% or less of your expected intake, your regular doctor will be notified.

If you are in the intervention group, the results from these food records will be given to you by a dietitian within 3 days after the collection of food records (Days 17, 31, and 45). You will receive these results in person with a dietitian consultant. You will be able to discuss any issues related to food intake (such as food choices, food options, problems related to meal preparation, and how to increase calories or nutrients) so that you might be able to bring up the caloric intake to good level.

You will be taken off this study if you develop a condition called gastrointestinal graft versus host disease, major organ failure (such as heart, kidney, or liver), or any intolerable side effects from the standard care treatment you are on.

This is an investigational study. Up to 12 patients will take part in this pilot study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has been diagnosed with cancer (leukemia or lymphoma).
2. Age 18 years or older
3. Subject has received their allogeneic BMT, fully ablative transplants, from either related or unrelated donors in the past 40 days
4. Subject can read, write, speak, and understand English
5. Subject has a caregiver (family member or friend) to keep the food diary record.
6. Subject voluntarily agrees and signs informed consent prior to participate in this study.
7. Subject is oriented to time, place, and person.

Exclusion Criteria:

1. Subject has major organ failure such as kidney, heart, or liver failure.
2. Subject has allergies to latex preventing use of the mouthpiece during indirect calorimetry testing.
3. Subject has been scheduled to withhold oral intake or parenteral nutrition support for more than 4 days during the week of dietary record (week 2, 4, and 6)
4. Subject has a diagnosis of gastro-intestinal graft versus host disease (GI-GVHD).
5. Subject has pre-transplant pulmonary function tests (PFTs) with force vital capacity (FVC) or forced expiratory volume in one second (FEV1) or diffusing capacity of the lung for carbon monoxide (DLCO) < 65% of predicted value.
6. Subject who is physically unable to complete the indirect calorimetry or who refuses calorimetry or who cannot understand the instructions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Patient Fatigue Scores <Brief Fatigue Inventory (BFI)> | BFI at study day 0, 14, 28, and 42

CONTACTS AND LOCATIONS:
Overall Officials: Srisuda Lecagoonporn, RN, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org